CLINICAL TRIAL: NCT01673191
Title: A 3-Month Clinical Trial to Assess the Safety and Efficacy of the OZURDEX® Intraocular Implant in Patients With Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Retinal Consultants of Arizona (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCA2012
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: Macular Edema; Diabetes Mellitus
MeSH Terms: conditions — Macular Edema; Diabetes Mellitus | interventions — Dexamethasone; Calcium Dobesilate; Steroids; Ketorolac; prednisolone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OZURDEX intraocular implant (Experimental): OZURDEX (dexamethasone posterior segment drug delivery system (DEX PS DDS), 0.7 mg
  Interventions: Drug: Dexamethasone intravitreal implant
- Steroid plus NSAID eye drop combination therapy (Active Comparator): NSAID eye drop: Acular LS Steriod eye drop: Pred Forte
  Interventions: Drug: Steroid plus NSAID eye drop combination therapy

INTERVENTIONS:
Drug: Dexamethasone intravitreal implant
  Other Names: OZURDEX
  Arms: OZURDEX intraocular implant
Drug: Steroid plus NSAID eye drop combination therapy
  Other Names: Acular LS and Pred Forte
  Arms: Steroid plus NSAID eye drop combination therapy

SUMMARY:
There is a need to find an effective therapy for diabetic patients who develop macular edema after cataract surgery.

DETAILED DESCRIPTION:
The objective of this study is to assess the safety and efficacy of the OZURDEX® intraocular implant in patients with diabetes mellitus, who develop macular edema after cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* Patient has diagnosis of Diabetes Mellitus, Type I or II.
* Patient has experienced the development of macular edema following cataract surgery in at least one eye.
* Patient has had cataract surgery within 90 days prior to the screening visit.

Exclusion Criteria:

* Patient has other significant ocular disease in study eye, including glaucoma.
* Patient has any active infection in the study eye.
* Patient has uncontrolled systemic illness (i.e., uncontrolled blood pressure, uncontrolled diabetes mellitus).
* Patient has experienced a significant increase in intraocular pressure following a prior treatment with topical or intravitreal steroidal medication.
* Patient has received the OZURDEX® implant before in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pravin U Dugel, MD, Principal Investigator — Retinal Consultants of Arizona
Locations (1):
- Retinal Consultants of Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- OZURDEX Intraocular Implant: OZURDEX (dexamethasone posterior segment drug delivery system (DEX PS DDS), 0.7 mg
  Dexamethasone intravitreal implant
- Steroid Plus NSAID Eye Drop Combination Therapy: NSAID eye drop: Acular LS Steriod eye drop: Pred Forte
  Steroid plus NSAID eye drop combination therapy
Period: Overall Study
Arm/Group | OZURDEX Intraocular Implant | Steroid Plus NSAID Eye Drop Combination Therapy
Started | 26 | 11
Completed | 26 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DEX IMPLANT ARM: Subects in the DEX implant arm received a single intravitreal administration of 0.7 mg OZURDEX in the study eye at the Day 0 appointment. In order to minimize subject discomfort, adequate local anesthesia was administered to the study eye prior to DEX implant injection. Immediately following DEX implant injection, the investigator performed indirect ophthalmic exam to assess for complications. In order to minimize risk of infection, a topical broad-spectrum antibiotic was placed in the study eye immediately prior to and following the injection, and the subject were provided a sample of a broad-spectrum antibiotic to use 4 times daily for 3 days following injection. The subject remained in the clinic for 15-30 minutes or until IOP <28 mmHg.
- Topical Steroid/NSAID ARM: Subjects randomized to receive the steroid/NSAID eye drop combination therapy began treatment at Day 0. The first administration occurred in clinic. Subjects was instructed how to instill eye drops properly and to instill each drop in the study eye four times per day every day until month 1 visit. At each monthly visit, subjects in this arm were assessed for the need to continue steroid/NSAID therapy.
- Total: Total of all reporting groups
Arm/Group | DEX IMPLANT ARM | Topical Steroid/NSAID ARM | Total
Number analyzed (Participants) | 26 | 11 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 4 | 16
  >=65 years | 14 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (7.6) | 68 (8.4) | 67.4 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 12 | 5 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 11 | 37
Best Corrected Visual Acuity [Mean (Standard Deviation); unit: logMAR units] — logMAR
  logMAR units | 0.49 (0.40) | 0.32 (0.22) | 0.44 (0.36)
Central Retinal Thickness [Mean (Standard Deviation); unit: micrometers] — Based on spectral domain optical coherence tomography (SD-OCT)
  micrometers | 402.2 (149.8) | 403.5 (156.2) | 402.5 (149.5)
Intraocular Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)] | 13.7 (2.8) | 14.4 (2.5) | 13.9 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Best Corrected Visual Acuity
Time Frame: 1 months
Measure: Mean (Standard Deviation); unit: logMAR units
Arm/Group | DEX IMPLANT ARM | Topical Steroid/NSAID ARM
Number analyzed (Participants) | 26 | 11
logMAR units | 0.3 (0.2) | 0.33 (0.37)

2. Primary Outcome: Mean Change in Best Corrected Visual Acuity
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: logMAR units
Arm/Group | DEX IMPLANT ARM | Topical Steroid/NSAID ARM
Number analyzed (Participants) | 26 | 11
logMAR units | 0.34 (0.46) | 0.22 (0.18)

3. Primary Outcome: Mean Change in Best Corrected Visual Acuity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR units
Arm/Group | DEX IMPLANT ARM | Topical Steroid/NSAID ARM
Number analyzed (Participants) | 26 | 11
logMAR units | 0.34 (0.45) | 0.21 (0.18)

4. Primary Outcome: Mean Change in Central Retinal Thickness
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | DEX IMPLANT ARM | Topical Steroid/NSAID ARM
Number analyzed (Participants) | 26 | 11
micrometers | 286.9 (66.1) | 360.8 (99.5)

5. Primary Outcome: Mean Change in Central Retinal Thickness
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | DEX IMPLANT ARM | Topical Steroid/NSAID ARM
Number analyzed (Participants) | 26 | 11
micrometers | 270.42 (46.8) | 336 (75.4)

6. Primary Outcome: Mean Change in Central Retinal Thickness
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | DEX IMPLANT ARM | Topical Steroid/NSAID ARM
Number analyzed (Participants) | 26 | 11
micrometers | 318.7 (103.2) | 341.1 (74.6)

7. Primary Outcome: Mean Change in Intraocular Pressure
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)
Arm/Group | DEX IMPLANT ARM | Topical Steroid/NSAID ARM
Number analyzed (Participants) | 26 | 11
millimeters of mercury (mm Hg) | 14.9 (3.3) | 14.1 (3)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | DEX IMPLANT ARM | Topical Steroid/NSAID ARM
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/11
Other Adverse Events (participants affected / at risk) | 1/26 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DEX IMPLANT ARM (N=26) | Topical Steroid/NSAID ARM (N=11)
Elevated Intraocular Pressure (Eye disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Limitations of our study include a small sample size and short-term follow up. Additional studies are needed to determine whether combination therapy with other treatments would be beneficial to patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No